CLINICAL TRIAL: NCT01951534
Title: Decisional Aid Intervention for Women Considering Breast Reconstruction
Acronym: BRDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 131025; R21CA149531-01A1 (NIH)
Record Dates: First submitted 2013-05-07; First posted 2013-09-26 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: breast reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breast Reconstruction Decisional Aid (BRDA) (Experimental): In the BRDA arm, participants will be provided with a website address for using the Breast Reconstruction Decisional Aid, a secure password, and instructions for using the website for the decisional aid.
  Interventions: Behavioral: Breast Reconstruction Decisional Aid (BRDA)
- Usual Care (UC) (Other): In the UC Condition, the participant will not be given the web-based decisional aid but will be given the Cancer Support Community pamphlet. This 56-page pamphlet contains information about the types of Breast Reconstruction, lists reasons why women choose reconstruction, key factors to considering when deciding, how to plan for surgery, possible risks, and a glossary of terms. The pamphlet is primarily informational. It is not customized, not interactive.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Breast Reconstruction Decisional Aid (BRDA)
  Arms: Breast Reconstruction Decisional Aid (BRDA)
Behavioral: Usual Care
  Arms: Usual Care (UC)

SUMMARY:
This is an intervention development and pilot study whose purpose is to determine the feasibility and acceptability of the breast reconstruction decisional aid (BRDA) and provide preliminary data on its impact on decisional outcomes.

The primary aim of this study is: "Is the intervention trial feasible?" The purpose is to develop a feasible web-based decisional aid (DA) for a larger scale trial. Thus it is important that this trial provide evidence of feasibility. The investigators will define feasibility as the rate of study acceptance and participation.

The secondary aim of this study is: " Is the BRDA acceptable and used?" The team will evaluate BRDA acceptability, use, difficulty with internet use, and what factors predict uptake and use. The investigators anticipate that, due to interest in the topic, the majority of women will access the website.

An additional secondary aim of this study is: "What is the impact of BRDA on BR knowledge, attitudes about BR, decisional conflict, preparedness and completeness of preparation, anxiety, and discussion with oncologist?" The purpose is to calculate effect sizes for a larger randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for a surgical consult with a breast surgeon
* Primary diagnosis of Stage 0 (Ductal Carcinoma in situ), 1, 2, or 3a breast cancer
* Patient speaks and reads English
* Patient is considering mastectomy

Exclusion Criteria:

* Patient who selects lumpectomy and not mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06-30 (Actual); Study Completion 2016-06-07 (Actual)

PRIMARY OUTCOMES:
Feasibility of a decisional aid to assist women with making the decision to undergo breast reconstruction | 3 years
  We will define feasibility as the rate of study acceptance and participation. First, we will examine acceptance as determined by consents and completed baselines. Second, we will examine time for completing surveys. We will judge this trial feasible if: 1) the acceptance rate among eligible patients is equal to or greater than 70%. We will judge completion rates at follow-up to be feasible for a larger scale trial if our completion rate is 75%. 2) If the survey length averages are > 35 minutes, we will deem this unacceptable and shorten the survey.

SECONDARY OUTCOMES:
Acceptability of BRDA | 3 years
  We will define acceptability using both quantitative and qualitative methods. Basic descriptive information will be automatically gathered from the DA tracking system regarding whether participants logged in, how many times, and for how long. Time spent in each module will be tracked and summarized. Participants will rate the DA and provide interview feedback regarding its ease of use. Interview feedback regarding home versus public access will be gathered. A second indicator of acceptability will be ratings on the DA evaluation and interview. The range of items on the scale is 1-7. An item mean of 4 is mid-range. We judge our intervention as acceptable if 75% of BRDA participants used the DA and if the average score on the evaluation was > 5.6, which is 80% of the highest score.
Impact of breast reconstruction decisional aid on knowledge and attitudes | 3 years
  This is an exploratory objective to calculate effect sizes for a larger randomized trial. Using survey data that we will collect as part of this research, we will look at the impact of BRDA on knowledge and attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Manne, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (9):
- United States (9):
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Southern Ocean Medical Center, Manahawkin, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania